CLINICAL TRIAL: NCT01155414
Title: Tolerance of Healthy Term Infants Fed Infant Formulas
Brief Title: Tolerance of Healthy Term Infants Fed Infant Formulas #4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK75
Record Dates: First submitted 2010-06-28; First posted 2010-07-01 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Term Infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Investigational infant formula A (Experimental): Investigational Protein Hydrolysate formula
  Interventions: Other: Investigational Infant Formula A
- Hydrolysate based Infant Formula (Active Comparator)
  Interventions: Other: Hydrolysate based infant formula
- Investigational Infant Formula B (Experimental): Investigational Protein Hydrolysate Formula
  Interventions: Other: Investigational Infant Formula B

INTERVENTIONS:
Other: Hydrolysate based infant formula — Infant formula ad lib
  Arms: Hydrolysate based Infant Formula
Other: Investigational Infant Formula A — Investigational infant formula ad lib
  Arms: Investigational infant formula A
Other: Investigational Infant Formula B — Investigational infant formula ad lib
  Arms: Investigational Infant Formula B

SUMMARY:
The primary objective of this study is to assess the comparative gastrointestinal (GI) tolerance of normal term infants to two experimental powdered formulas compared with a commercially available powdered formula.

ELIGIBILITY:
Inclusion Criteria:

* Singleton full term birth in good health
* Birth weight was > 2490 g.
* Between 0 and 8 days of age.
* Infants using medications (including OTC such as Mylicon® for gas), home remedies (such as juice for constipation), herbal preparations or rehydration fluids that might affect GI tolerance may not be enrolled unless both the parent and the physician agree to discontinue these agents prior to enrollment.
* Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study, unless instructed otherwise by their healthcare professional.
* Parent(s) confirm their intention not to administer vitamin or mineral supplements, solid foods or juices to their infant from enrollment through the duration of the study.

Exclusion Criteria:

• An adverse maternal, fetal or infant medical history and treatment with antibiotics

Ages: 1 Day to 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
GI tolerance via stool consistency | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, PhD, Study Chair — Abbott Nutrition
Locations (10):
- United States (10):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Dothan, Alabama
  - SCORE Physician Alliance, St. Petersburg, Florida
  - University of Iowa, Coralville, Iowa
  - Medical Associates Clinic, PC, Dubuque, Iowa
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio Pediatric Research Association, Huber Heights, Ohio
  - Institute of Clinical Research, Mayfield Heights, Ohio
  - Pediatric Clinical Research Office, Hershey, Pennsylvania
  - The Jackson Clinic, PA, Jackson, Tennessee